CLINICAL TRIAL: NCT03334214
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability and Pharmacodynamics of ISIS 484137 (IONIS-DGAT2Rx, an Antisense Inhibitor of Diacylglycerol Acyltransferase 2) Administered Once-Weekly for 13 Weeks in Adult Patients With Type 2 Diabetes
Brief Title: Safety, Tolerability, and Pharmacodynamics of IONIS-DGAT2Rx in Adult Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 484137-CS2; 2017-003197-13 (EudraCT Number)
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatic Steatosis
Keywords: Hepatic Steatosis; IONIS-DGAT2Rx; Type 2 Diabetes
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IONIS DGAT2Rx (Experimental): Single Dose of DGAT2Rx administered subcutaneously once weekly for 13 weeks
  Interventions: Drug: IONIS DGAT2Rx
- Placebo (sterile saline 0.9) (Placebo Comparator): Calculated volume to match active comparator administered subcutaneously once weekly for 13 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS DGAT2Rx — Single Dose of DGAT2Rx administered subcutaneously once weekly for 13 weeks
  Arms: IONIS DGAT2Rx
Drug: Placebo — Saline 0.9%
  Arms: Placebo (sterile saline 0.9)

SUMMARY:
The purpose is to assess the Safety, Tolerability, and Pharmacodynamics effect of IONIS DGAT2Rx in up to 45 Adult Patients with Type 2 Diabetes.

DETAILED DESCRIPTION:
This short-term study will assess changes in hepatic steatosis over a 13-week treatment period in a patient population with higher risk for development of Nonalcoholic fatty liver disease (NAFLD) and Nonalcoholic steatohepatitis (NASH), obese type 2 diabetes mellitus (T2DM) with elevated HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements.
* Males or females aged 18-75, inclusive, at the time of Informed Consent.
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal.
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method.
* Body mass index (BMI) ≥ 27.0 - ≤ 39.0 kilograms per square meter (kg/m^2).
* Diagnosis of Type 2 Diabetes Mellitus with an Hemoglobin A1C (HbA1c) ≥7.3% and ≤9.5% at screening.
* Must have been on a stable dose of Oral Antidiabetic Therapy for a minimum of 3 months prior to Screening.
* ≥ 10% liver fat prior to randomization assessed by MRI-PDFF.
* Stable body weight for at least 3 months before screening.

Exclusion Criteria:

* Clinically-significant abnormalities in medical history or physical examination.
* Clinically-significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion, per Sponsor.
* Evidence of uncorrected hypothyroidism or hyperthyroidism results at Screening.
* History of solid organ transplantation or renal dialysis.
* Clinically-significant complications of diabetes.
* Treatment with another Study Drug, biological agent, or device within one-month of screening.
* Known history or evidence of liver disease with a positive test for human immunodeficiency virus (HIV), Hepatitis C virus (HCV), or chronic Hepatitis B virus (HBV), or chronic liver disease other than NASH.
* Recent history of, or current drug or alcohol abuse.
* Current use of concomitant medications known to significantly impact body weight or that may cause liver toxicity, per Investigator
* Use of anticoagulant/Antiplatelet agents unless the dose has been stable for 4 weeks prior to the first dose of study drug]
* Use of non-steroidal anti-inflammatory drug nimesulide or any other drug influencing coagulation (except lose-dose aspirin).
* Use of obeticholic acid or ursodeoxycholic acid
* Considered unsuitable for inclusion by the Principal Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Bhanot, Study Director — Ionis Pharmaceuticals, Inc.
Locations (17):
- Canada (2):
  - Ionis Investigational Site, Halifax, Nova Scotia
  - Ionis Investigational Site, Chicoutimi, Quebec
- Hungary (4):
  - Ionis Investigational Site, Budapest
  - Ionis Investigational Site, Hatvan
  - Ionis Investigational Site, Miskolc
  - Ionis Investigational Site, Székesfehérvár
- Poland (9):
  - Ionis Investigational Site, Bydgoszcz
  - Ionis Investigational Site, Bytom
  - Ionis Investigational Site, Chełm
  - Ionis Investigational Site, Katowice
  - Ionis Investigational Site, Krakow
  - Ionis Investigational Site, Lodz
  - Ionis Investigational Site, Mysłowice
  - Ionis Investigational Site, Wierzchosławice
  - Ionis Investigational Site, Wroclaw
- United Kingdom (2):
  - Ionis Investigational Site, Dundee
  - Ionis Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loomba R, Morgan E, Watts L, Xia S, Hannan LA, Geary RS, Baker BF, Bhanot S. Novel antisense inhibition of diacylglycerol O-acyltransferase 2 for treatment of non-alcoholic fatty liver disease: a multicentre, double-blind, randomised, placebo-controlled phase 2 trial. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):829-838. doi: 10.1016/S2468-1253(20)30186-2. Epub 2020 Jun 15. PMID 32553151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 participants were randomized at multiple study centers in Canada, Hungary, and Poland.
Pre-assignment Details: A total of 173 participants were screened for the study and 44 participants were randomized and received study drug.
Groups:
- Placebo: Calculated volume to match active comparator administered subcutaneously once weekly for 13 weeks.
- IONIS DGAT2Rx 250 mg: Single dose of DGAT2Rx administered subcutaneously once weekly for 13 weeks.
Period: Overall Study
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Started | 15 | 29
Completed | 14 | 27
Not Completed | 1 | 2
Not completed — Adverse Event or Serious Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Population: All subjects who are randomized into the study regardless of whether they received Study Drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg | Total
Number analyzed (Participants) | 15 | 29 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6) | 62 (7) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 29 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 29 | 44
Liver Fat Percentage (Randomized Population) [Mean (Standard Deviation); unit: fat percentage] | 19.54 (5.68) | 18.48 (6.04) | 18.84 (5.88)
Liver Fat Percentage (Per Protocol Population) [Mean (Standard Deviation); unit: fat percentage] — Population: The per protocol set included all randomized participants who received at least 10 of the prescribed doses and received the first 4 doses in the first 5 weeks, not missing 3 consecutive weekly doses and having no significant protocol deviations.
  fat percentage
    number analyzed (Participants) | 12 | 25 | 37
    (all) | 19.77 (6.03) | 18.22 (6.05) | 18.72 (6.00)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Liver Fat Percentage (Randomized Population)
Description: Absolute change in liver fat percentage as quantified by magnetic resonance imaging-estimated proton density fat fraction (MRI-PDFF) from baseline to post-treatment MRI.
Time Frame: Baseline to Week 15
Population: The randomized population included all participants who are randomized into the study regardless of whether they received the study drug.
Measure: Mean (Standard Deviation); unit: liver fat percentage
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 15 | 26
liver fat percentage | -0.04 (5.82) | -5.37 (5.41)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.003, ANOVA

2. Primary Outcome: Absolute Change in Liver Fat Percentage (Per Protocol Population)
Description: Absolute change in liver fat percentage as quantified by MRI-PDFF from baseline to post-treatment MRI.
Time Frame: Baseline to Week 15
Population: The per protocol set included all randomized participants who received at least 10 of the prescribed doses and received the first 4 doses in the first 5 weeks, not missing 3 consecutive weekly doses and having no significant protocol deviations.
Measure: Mean (Standard Deviation); unit: liver fat percentage
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
liver fat percentage | -0.64 (6.11) | -5.15 (5.40)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.026, ANOVA

3. Primary Outcome: Percentage of Participants With Adverse Events That Were Related to Treatment With IONIS DGAT2Rx
Description: An adverse event (AE) is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.
Time Frame: Up to 176 days
Population: The safety set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 15 | 29
percentage of participants | 13.3 | 48.3

4. Primary Outcome: Percentage of Participants With Adverse Events, Graded by Severity, That Were Related to Treatment With IONIS DGAT2Rx
Description: AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010. Grades: mild - the event is easily tolerated by the participant and does not affect the participant's usual daily activities; moderate - the event causes the participant more discomfort and interrupts the participant's usual daily activities; severe - the event is incapacitating and causes considerable interference with the participant's usual daily activities.
Time Frame: Up to 176 days
Population: The safety set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 15 | 29
percentage of participants
  Mild | 6.7 | 37.9
  Moderate | 6.7 | 6.9
  Severe | 0.0 | 3.4

5. Secondary Outcome: Percent Change in Liver Fat Percentage
Description: Relative percent change in liver fat percentage from baseline to post-treatment MRI.
Time Frame: Baseline to Week 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percent change | -2.4 (28.8) | -25.5 (26.5)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.024, ANOVA

6. Secondary Outcome: Percentage of Participants With ≥ 30% Relative Reduction in Liver Fat Percentage
Description: Percentage of participants with ≥ 30% relative reduction in liver fat percentage from baseline to post-treatment.
Time Frame: Week 15
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percentage of participants | 16.7 | 48.0
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.0774, Cochran-Mantel-Haenszel; The p-value is obtained using Cochran-Mantel-Haenszel (CMH) test stratified by the baseline liver fat stratum (<20%, ≥20%) stratification factor

7. Secondary Outcome: Percent Change in Liver Volume
Description: Assessed from Baseline MRI to Post-Treatment MRI.
Time Frame: Baseline to Week 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percent change | -1.9 (7.2) | -6.3 (9.8)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.183, ANOVA

8. Secondary Outcome: Percent Change in Plasma Lipoprotein Profile
Description: Percent change in plasma lipoprotein profile (total cholesterol, apolipoprotein B [ApoB], high density lipoprotein (HDL), low density lipoprotein cholesterol [LDL-C], non-HDL, triglycerides, and very low density lipoproteins [VLDL]) from baseline to the average of the post-treatment values assessed 1 and 2 weeks after the last dose (Post-Treatment 1 and Post-Treatment 2 visits).
Time Frame: Week 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percent change
  Total cholesterol | -4.4 (9.6) | -2.9 (14.2)
  ApoB | -8.1 (9.5) | -6.7 (15.3)
  HDL | 1.0 (6.3) | 2.2 (11.6)
  LDL-C | -8.8 (14.9) | -3.8 (24.1)
  Non-HDL | -7.1 (13.4) | -3.8 (18.7)
  Triglycerides | -0.8 (20.3) | 2.8 (20.1)
  VLDL-C | -0.7 (20.3) | 2.0 (18.5)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Total Cholesterol; Test type: Superiority; p = 0.682, ANOVA
Statistical Analysis 2: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; ApoB; Test type: Superiority; p = 0.716, ANOVA
Statistical Analysis 3: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; HDL; Test type: Superiority; p = 0.717, ANOVA
Statistical Analysis 4: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; LDL-C; Test type: Superiority; p = 0.463, ANOVA
Statistical Analysis 5: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Non-HDL; Test type: Superiority; p = 0.555, ANOVA
Statistical Analysis 6: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Triglycerides; Test type: Superiority; p = 0.619, ANOVA
Statistical Analysis 7: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; VLDL-C; Test type: Superiority; p = 0.698, ANOVA

9. Secondary Outcome: Percent Change in Parameters of Insulin Resistance (IR)
Description: Percent change in parameters of IR (fasting plasma glucose [FPG], homeostatic model assessment - insulin resistance [HOMA-IR], and insulin) from baseline to post-treatment.
Time Frame: Week 14
Population: The per protocol set included all randomized participants who received at least 10 of the prescribed doses and received the first 4 doses in the first 5 weeks, not missing 3 consecutive weekly doses and having no significant protocol deviations. Number analyzed were the participants with analysis values at specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percent change
  FPG: number analyzed (Participants) | 12 | 24
  FPG | -6.3 (23.1) | -6.9 (16.1)
  HOMA-IR: number analyzed (Participants) | 12 | 24
  HOMA-IR | -16.9 (29.7) | 2.6 (46.8)
  Insulin: number analyzed (Participants) | 12 | 24
  Insulin | -10.3 (21.7) | 10.1 (44.8)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; FPG; Test type: Superiority; p = 0.902, ANOVA
Statistical Analysis 2: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; HOMA-IR; Test type: Superiority; p = 0.267, Van Elteren test
Statistical Analysis 3: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Insulin; Test type: Superiority; p = 0.200, Van Elteren test

10. Secondary Outcome: Absolute Change in Hemoglobin A1C (HbA1C)
Description: Absolute change in HbA1C from baseline to post-treatment.
Time Frame: Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
Number analyzed (Participants) | 12 | 25
percentage of total hemoglobin | -0.2 (0.7) | -0.2 (0.6)
Statistical Analysis 1: Comparison: Placebo vs IONIS DGAT2Rx 250 mg; Test type: Superiority; p = 0.933, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 176 days
Description: The safety set included all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | IONIS DGAT2Rx 250 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/15 | 4/29
Other Adverse Events (participants affected / at risk) | 10/15 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | IONIS DGAT2Rx 250 mg (N=29)
Cardiac arrest (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | IONIS DGAT2Rx 250 mg (N=29)
Injection site erythema (General disorders) | 0 | 10
Injection site bruising (General disorders) | 1 | 4
Injection site swelling (General disorders) | 0 | 5
Injection site pain (General disorders) | 0 | 4
Injection site pruritus (General disorders) | 0 | 4
Fatigue (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03334214/Prot_SAP_000.pdf